CLINICAL TRIAL: NCT02664974
Title: Home Enteral Nutrition in Malnourished Patients With Gastrointestinal Cancer: A Multicenter Randomized Clinical Trial
Brief Title: Home Enteral Nutrition in Malnourished Patients With Gastrointestinal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HEN
Record Dates: First submitted 2016-01-13; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Malnutrition; Gastrointestinal Cancer
MeSH Terms: conditions — Malnutrition; Gastrointestinal Neoplasms | interventions — Enteral Nutrition; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HEN group (Experimental): Home Enteral Nutrition
  Interventions: Dietary Supplement: Enteral nutrition
- Control group (Active Comparator): Dietary Counseling
  Interventions: Other: Dietary counseling

INTERVENTIONS:
Dietary Supplement: Enteral nutrition — Home Enteral Nutrition was planned to cover the basal energy requirement calculated with Harris Benedict Formula, it was administrated preferentially during nocturnal hours as an integration of oral diet.
  Enteral Nutrition included any standard polymeric formula providing 1-1.5 Kcal/mL with carbohydrates 50%-60%, lipids 25%-35% and protein 12%-20%.
  Home Enteral Nutrition can be withdrawn in the treated group, after 2 months from discharge, whenever a weight gain ≥ 5% is reported, and oral alimentation is regular and adequate.
  Arms: HEN group
Other: Dietary counseling — Specific nutritional advices including total energy and protein requirements were provided to patients and oral high-calorie supplements were prescribed whenever necessary.
  Home Enteral Nutrition can be started in patients of the control group, not before two months from discharge, if a further weight loss ≥ than 5% is reported.
  Arms: Control group

SUMMARY:
Phase III, medical, multicentric, controlled, open label, two-parallel groups, randomized, clinical trial.

The aim of this study is to evaluate the efficacy of home enteral nutrition on the nutritional status, the quality of life and tolerance to chemotherapy, in malnourished patients who undergo major gastrointestinal surgery for malignancy (oesophagus, stomach, pancreas, biliary tract). Patients were randomized to receive either home enteral nutrition (HEN, treatment group) or nutritional counselling (control group).

ELIGIBILITY:
Inclusion Criteria:

* Both gender with age higher than 18 years.
* Documented cancer of the gastrointestinal tract: oesophagus, stomach, pancreas, biliary tract
* Candidate for major elective surgery.
* Preoperative nutritional risk score ≥ 3
* Written informed consent.

Exclusion Criteria:

* Age < 18 years
* Karnofsky index < 60
* Renal insufficiency (Ongoing haemodialysis or plasma creatinine > 3 mg/dL)
* Respiratory insufficiency
* Child-Pugh class C
* Short Bowel Syndrome
* Pregnancy
* Emergency operation
* Foreign residence or residence in Italian region with no regulation designed for home artificial nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maintenance of body weight | 2 months
  Evaluated by weight change after discharge

SECONDARY OUTCOMES:
Improvement of quality of life | 2 months
  Evaluated at hospital admission and two months after discharge by the self-administrated Functional Assessment of Anorexia/Cachexia Therapy (FAACT) questionnaire
Improvement of tolerance to chemotherapy | 6 months
  Evaluated by the ratio chemotherapy planned / chemotherapy administered

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Gavazzi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (2):
- Italy (2):
  - European Institute of Oncology, Milan, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan